CLINICAL TRIAL: NCT06340763
Title: JET Enhanced Thrombectomy Intervention Hong Kong Post Market Study
Brief Title: JETi Hong Kong Post Market Study (PMS)
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10466; CRD_1058 (Other: Abbott)
Record Dates: First submitted 2024-03-12; First posted 2024-04-01 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Venous Thrombosis; Peripheral Arterial Thrombosis; Peripheral Arteriovenous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- JETi Hydrodynamic Thrombectomy System: Subject was treated or is expected to be treated for acute/subacute thrombosis in the peripheral vasculature with the JETi Hydrodynamic Thrombectomy System.
  Interventions: Device: JETi Hydrodynamic Thrombectomy System

INTERVENTIONS:
Device: JETi Hydrodynamic Thrombectomy System — The JETi Hydrodynamic Thrombectomy System is a hydro-mechanical aspiration system intended for the removal of intravascular thrombus. The system is comprised of the JETi Catheter, JETi Pump Set, and JETi Saline Drive Unit (SDU), accessory cart, suction tubing, and non-sterile canister set. The JETi System is designed to simultaneously deliver a stream of high-pressure saline via a displacement pump to the distal tip of the JETi Catheter, while aspirating thrombotic material macerated by the saline stream.

SUMMARY:
The JETi Hong Kong PMS is a single-arm, multicenter study to collect real-world data on the safety, performance, and clinical benefits of the JETi System for the treatment of acute and subacute thrombosis in the peripheral vasculature. This is a post-market study that will register approximately 20 subjects at approximately 5 centers in Hong Kong. Subjects participating in this study will be followed for up to 30 days (in cases of prospective consent) after Day 0. Day 0 is defined as the day when the JETi catheter is introduced into the intended vasculature of the subject.

DETAILED DESCRIPTION:
The JETi System is a hydro-mechanical aspiration system manufactured by Abbott Medical, consisting of a catheter, pump set, and accessories. The system is intended to remove/aspirate fluid and break-up soft emboli and thrombus from the peripheral vasculature and to subselectively infuse/deliver diagnostics or therapeutics with or without vessel occlusion.

This study will collect data on how the JETi System performs in the treatment of patients undergoing a percutaneous thrombectomy procedure for peripheral thrombosis. Subjects treated for arterial, venous, or arteriovenous thromboses, and subject with diagnoses such as acute limb ischemia (ALI), chronic limb ischemia/chronic limb threatening ischemia (CLI/CTLI), peripheral artery disease (PAD), deep vein thrombosis (DVT), hemodialysis access thrombosis, and others may be included.

Both prospective and retrospective consent (if all assessments needed for the primary endpoints are complete) are permitted. After index procedure, subjects will be evaluated at discharge and 30 days in cases of prospective consent. In cases of retrospective consent, duration of participation will vary. If consent occurs after the procedure and prior to 30 days, the subject will be asked to return for a 30-day visit. If consent occurs after 30 days, the subject will not need to return for a study visit. Relevant data will be collected from the medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Subject was treated or is expected to be treated for acute/subacute thrombosis, as determined by investigator, in the peripheral vasculature with the JETi Hydrodynamic Thrombectomy System.
2. Subject or legally authorized representative must provide written informed consent
3. Subject must be ≥ 18 years of age and of Asian race.

Exclusion Criteria:

1. Subject has previously been registered in the JETi Hong Kong PMS in the last 12 months unless treated in the contralateral limb/different anatomy; patients treated in the contralateral limb/different anatomy within the last 12 months may re-enroll in the study.
2. Subject is currently participating in another drug or device clinical investigation.
3. Subject has active symptoms and/or a positive test result of COVID-19 or other rapidly spreading infectious agent within the past 20 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects of all genders from the patient population undergoing percutaneous treatment of thrombosis in the peripheral vascular system will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Hong Kong (4):
  - Princess Margaret Hospital, Hong Kong, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong, Hong Kong
  - Queen Mary Hospital, Hong Kong, Hong Kong
  - Prince of Wales Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 subjects were registered in the JETi Hong Kong PMS across 3 sites in Hong Kong between August 7, 2024 and January 24, 2025.
Period: Overall Study
Arm/Group | JETi Hydrodynamic Thrombectomy System
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | JETi Hydrodynamic Thrombectomy System
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Year] | 68.9 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Intended Vasculature [Count of Participants; unit: Participants]
  Artery | 7
  Vein | 2
  Arteriovenous | 3
Diagnosis [Count of Participants; unit: Participants]
  Acute Limb Ischemia | 6
  Peripheral Artery Disease with Claudication (Rutherford 1-3) | 1
  Hemodialysis Access: AV Fistula Thrombosis | 2
  Hemodialysis Access: AV Graft Thrombosis | 1
  Deep Vein Thrombosis | 2

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint - For Arterial and Arteriovenous Subjects: Clot Removal Grade for Each JETi-treated Vessel
Description: Clot removal grade for each JETi-treated target vessel from pre-JETi angiogram to post-JETi angiogram (post-JETi thrombectomy and prior to any adjunctive therapies to treat underlying culprit lesions) per the grades (vessel basis). The independent imaging core laboratory will be responsible for assessing this endpoint.
  The rate of clot removal grade for each JETi-treated target vessel will be measured as per the Grades below:
  Grade I: < 50% reduction; Grade II: 50- <95% reduction; Grade III: 95-100% reduction.
Time Frame: During the procedure
Population: The number of participants analyzed includes arterial and arteriovenous subjects who had available data.
Measure: Count of Units; unit: Vessels
Units Other Than Participants: Vessels
Groups:
- JETi Hydrodynamic Thrombectomy System: Subject was treated or is expected to be treated for arterial or arteriovenous thrombosis with the JETi Hydrodynamic Thrombectomy System.
  JETi Hydrodynamic Thrombectomy System: The JETi Hydrodynamic Thrombectomy System is a hydro-mechanical aspiration system intended for the removal of intravascular thrombus. The system is comprised of the JETi Catheter, JETi Pump Set, and JETi Saline Drive Unit (SDU), accessory cart, suction tubing, and non-sterile canister set. The JETi System is designed to simultaneously deliver a stream of high-pressure saline via a displacement pump to the distal tip of the JETi Catheter, while aspirating thrombotic material macerated by the saline stream.
Arm/Group | JETi Hydrodynamic Thrombectomy System
Number analyzed (Participants) | 9
Number analyzed (Vessels) | 9
Vessels
  Grade I | 2
  Grade II | 2
  Grade III | 5

2. Primary Outcome: Primary Safety Endpoint - For Arterial and Arteriovenous Subjects: Composite of JETi-related Major Adverse Events (MAEs)
Description: JETi-related major adverse events (MAEs), defined as the following JETi-related events adjudicated by a clinical events committee (CEC) (subject basis): death, major amputation of the treated limb, or major bleeding.
Time Frame: Up to 30 days post-index procedure
Population: The number of participants analyzed includes arterial and arteriovenous subjects who had available data.
Measure: Number; unit: Participants
Groups:
- JETi Hydrodynamic Thrombectomy System: Subject was treated or is expected to be treated for arterial or arteriovenous thrombosis with the JETi Hydrodynamic Thrombectomy System.
Arm/Group | JETi Hydrodynamic Thrombectomy System
Number analyzed (Participants) | 10
Participants | 0

3. Primary Outcome: Primary Effectiveness Endpoint - For Venous Subjects: Percent of Treated Vessel(s) With ≥ 75% Venous Thrombus Reduction Via Modified Marder Score (Limb Basis).
Description: Percent of treated vessel(s) with ≥ 75% venous thrombus reduction from pre-JETi venogram to final venogram (post-JETi AND after any/all adjunctive therapies to treat underlying culprit lesions) via modified Marder score (limb basis). If no adjunctive therapies or devices are used after JETi, post-JETi score is also final score.
Time Frame: During the procedure
Population: The number of participants analyzed includes venous subjects who had available data.
Measure: Count of Units; unit: Vessels
Units Other Than Participants: Vessels
Groups:
- JETi Hydrodynamic Thrombectomy System: Subject was treated or is expected to be treated for lower extremity DVT with the JETi Hydrodynamic Thrombectomy System.
Arm/Group | JETi Hydrodynamic Thrombectomy System
Number analyzed (Participants) | 2
Number analyzed (Vessels) | 2
Vessels | 1

4. Primary Outcome: Primary Safety Endpoint - For Venous Subjects: Composite of JETi-related Major Adverse Events (MAEs)
Description: JETi-related major adverse events (MAEs), defined as the following JETi-related events adjudicated by a clinical events committee (CEC): death, symptomatic pulmonary embolism (PE), major bleeding, or re-thrombosis of JETi-treated vessel(s).
Time Frame: Up to 30 days post-index procedure
Population: The number of participants analyzed includes venous subjects who had available data.
Measure: Number; unit: Participants
Arm/Group | JETi Hydrodynamic Thrombectomy System
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 30 days
Arm/Group | JETi Hydrodynamic Thrombectomy System
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JETi Hydrodynamic Thrombectomy System (N=12)
Endocarditis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT06340763/Prot_SAP_000.pdf